CLINICAL TRIAL: NCT04944927
Title: Role of Alternating Hemiplegia of Childhood Genotype in Cardiac Repolarization. HEART: HEmiplegia Arrhythmia Retrospective Trial
Brief Title: HEmiplegia Arrhythmia Retrospective Trial
Acronym: HEART
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0493
Record Dates: First submitted 2021-06-02; First posted 2021-06-30 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Alternating Hemiplegia of Childhood
Keywords: QTc; Cardiac repolarization and arrhythmia; ECG; Alternating Hemiplegia
MeSH Terms: conditions — Alternating hemiplegia of childhood; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Alternating Hemiplegia of Childhood: Patients that meet the clinical diagnostic criteria (Aicardi et al, 1995) for typical alternating hemiplegia with or without identified mutations in ATP1A3.
  At least one prolonged ECG study available is required.
  Interventions: Other: Recording of clinical parameters and electrocardiogram parameters

INTERVENTIONS:
Other: Recording of clinical parameters and electrocardiogram parameters — Retrospective recording of demographic information (age, sex, age at diagnosis), genetic information, cardiological information, pharmacological treatments, electrocardiogram data. All above data will be deidentified.

SUMMARY:
Alternating Hemiplegia of Childhood (AHC) is a rare and severe disease that is in need of effective, and hopefully even curative, therapies. Afflicted patients suffer from severe paralyzing crises, often excruciatingly painful muscle spasms, severe often life threatening epileptic seizures, frequently severe developmental and psychiatric/psychological disabilities and other comorbidities, such as cardiac disturbances. Recent data indicate that AHC genotype is in relation to cardiac repolarization troubles and to cardiac arrhythmias. The primary hypothesis to explore is that there is an association between genotype and cardiac phenotype in AHC.

ELIGIBILITY:
Inclusion Criteria:

* Patients that meet the clinical diagnostic criteria (Aicardi et al, 1995) for typical alternating hemiplegia with or without identified mutations in ATP1A3.
* At least one ECG study is required.
* Patients ages yearand more

Exclusion Criteria:

* Informed consent or assent not obtainable
* ATP1A3 testing not performed
* No ECG studies are available

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Alternating Hemiplegia of Childhood
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Measurement of QTc interval and all relevant cardiac repolarization measurements | Day 1
  Outcome measure: QTc interval and cardiac repolarization measurement in milliseconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Epileptology, Sleep Disorders and Functional Neurology in Children, Hôpital Femme Mère Enfant, University Hospitals of Lyon (Hospices Civils de Lyon), Bron, France